CLINICAL TRIAL: NCT03115125
Title: Descriptive Study of the Evolution in Proportion of Regulatory B Lymphocytes in Patients Hospitalized in Intensive Care for Severe Sepsis
Acronym: DELyBREG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2015_843_0028
Record Dates: First submitted 2017-04-04; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Severe Sepsis
Keywords: B lymphocyte
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients with severe sepsis (Other)
  Interventions: Other: Describe for the first time the kinetics of evolution in proportion of the circulating Brég in patients with severe septic state, at times D0, D2, D7 and D14 of hospitalization in medical reanimation.

INTERVENTIONS:
Other: Describe for the first time the kinetics of evolution in proportion of the circulating Brég in patients with severe septic state, at times D0, D2, D7 and D14 of hospitalization in medical reanimation. — Describe for the first time the kinetics of evolution in proportion of the circulating Brég in patients with severe septic state, at times D0, D2, D7 and D14 (or on leaving the service if before D14) of hospitalization in medical reanimation.

SUMMARY:
Severe sepsis and septic shock are the most severe forms of sepsis (which associates a systemic inflammatory response with infection). These are serious pathologies with a lethality estimated at almost 40% at 28 days (after the onset of sepsis).

After a first pro-inflammatory phase, a second compensatory phase called Compensatory Anti-Inflammatory Response Syndrome (CARS) takes place quickly. Patients then show signs of immunosuppression and profound alterations in immune functions. It is during this phase that the vast majority of deaths occur, far from the onset of the shock, which is related to the inability of the immune system to eliminate the initial infectious agent and / or a greater susceptibility Important to develop secondary infections (nosocomial infection, latent virus reactivation ...).

The CARS phase has been the subject of studies focusing on measuring the plasma concentration of anti-inflammatory cytokines (such as Interleukin (IL) -10), the percentage of regulatory T lymphocytes (Treg), Or the percentage of monocytic expression of HLA-DR in septic patients.

The investigator proposes to carry out the first study on a newly described regulatory lymphocytic subpopulation: regulatory B lymphocytes (Breg) from a quantitative and functional point of view in severe septic states.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with severe sepsis or septic shock diagnosed less than 24 hours (defined as D0) and hospitalized in the medical resuscitation department of the Amiens-Picardie University Hospital.
* The definitions of severe sepsis and septic shock are the result of the consensus of the Société de Réanimation de Langue Française dating from 2005:

  * Sepsis refers to a systemic inflammatory response syndrome (SIRS) in the presence of suspected or identified infection. Sepsis is said to be severe when lactate> 4 mmol / L or arterial hypotension prior to filling or organ dysfunction is present (one is sufficient): hypoxemia with a PaO2 / FIO2 <300 ratio, renal failure with Hepatic insufficiency with INR> 4 or bilirubin> 78 μmol / l, thrombocytopenia (platelets <100 000 / mm3) and hepatic insufficiency> 176 μmol / l, coagulation disorders with INR> 1.5 Disorders of higher functions with a Glasgow Coma Score <13.
  * Finally, septic shock is defined as a severe sepsis condition with persistent hypotension despite a well-conducted vascular filling (20-40 ml / kg isotonic saline).

Exclusion Criteria:

* Patient with active neoplasia, immune deficiency, autoimmune disease or autoimmune disease.
* Patient under tutorship or curatorship
* Taking an immunomodulatory or immunosuppressive treatment at the time of the study or the year prior to hospitalization for sepsis.
* Antecedent or haematopoietic graft in progress.
* Pregnancy in progress.
* Known history of infection with human immunodeficiency virus (HIV) type 1 or 2 or with hepatitis B or C virus
* Patient with agranulocytosis (defined as neutrophils <0.5 G / L).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04-20 (Actual); Primary Completion 2017-05-19 (Estimated); Study Completion 2017-05-19 (Estimated)

PRIMARY OUTCOMES:
Variation in the proportion of circulating Breg compared to total B lymphocytes in the included cohort of patients | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France